CLINICAL TRIAL: NCT06234670
Title: Risk Factors and A Prediction Model of Recurrence of Uterine Fibroids
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Wenwen Wang (Other)
Collaborators: Tongji Hospital (Other)
Responsible Party: Sponsor-Investigator, Wenwen Wang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: V1.0
Record Dates: First submitted 2023-12-21; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Uterine Fibroid; Recurrence
Keywords: Uterine Fibroid; Recurrence; Risk factor; Prediction medel
MeSH Terms: conditions — Leiomyoma; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with uterine fibroids accepted myomectomy.: Complete the observation and follow-up, to identify the outcome （recur or not recur).
  Interventions: Other: No intervertion

INTERVENTIONS:
Other: No intervertion — This study is a retrospective observational study without intervention.

SUMMARY:
To research risk factors for recurrence of uterine fibroids and build a prediction model of recurrence of uterine fibroids to facilitate the early detection as well as the early intervention for patients who are prone to recur.

DETAILED DESCRIPTION:
Uterine fibroids are the most common benign tumors of female reproductive organs during childbearing age. With the emphasis on fertility preservation and the pursuit of the physical integrity, about 46% of patients prefer the conservative surgery which preserves the uterus. However, the high recurrence rate of uterine fibroids after conservative surgery does cause formidable clinical problems.

According to the literature, the recurrence rate is about 11.7% at one year after myomectomy and would increase steadily. At the eighth year of myomectomy, the recurrence rate is as high as 84.4%. During the long-term follow-up, about one-third of patients eventually require reoperation.

Recurrence not only leads to the recurrence of fibroid-related symptoms such as anemia, abdominal and pelvic pain, frequent urination and urgency, abnormal stool, etc., but also increases the burden of economic and national medical insurance, besides, it even causes serious problems such as psychological disorders, infertility, adverse pregnancy outcomes and malignant transformation, which affecting physical and mental health as well as destroying family happiness and threatening national population security.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-50 years
2. Diagnosed with uterine fibroids （by ultrasound or pathology）
3. Accept myomectomy.
4. Complete clinical data.

Exclusion Criteria:

1. Severe infectious disease
2. Previous history of malignant tumors
3. Incomplete clinical data.
4. Pregnant

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female patients with uterine fibroids
Study Population: Female patients with uterine fibroids and accept myomectomy.
Sampling Method: Probability Sample
Enrollment: 3200 (Estimated)
Dates: Start 2024-01-25 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
The performance of the prediction model for recurrence of uterine fibroids as assessed by AUC | through study completion, about June.2025
  Complete the follow-up, and compare the actual recurrence population with the predicted recurrence population to judge the performance of the prediction model. Use the AUC (Area Under Curve)

SECONDARY OUTCOMES:
Numbers of risk factors of recurrent uterine fibroids as certained by statistic analysis | about June.2024
  To identify the risk factors of recurrent uterine fibroids. We identify the risk factors through statistic analysis. Statistical significance proves to be the symbol of identifycation of risk factors.
The recurrence rate of uterine fibroids yearly | about Febrary.2024
  To calculate the recurrence rate of uterine fibroids yearly
The fertility rate after myomectomy | about Febrary.2024
  To research the fertility rate after myomectomy and evaluate the impact of the surgery.
The quality of life after myomectomy will be assessed by UFS-QOL,(uterine fibroid symptom and health-related quality of life, UFS-QOL) | through study completion, about June.2025
  To assess the quality of life after myomectomy, we use UFS-QOL.The UFS-QOL, the most popular self-administered instrument in assessing the whole spectrum of fibroid-related symptoms and health-related quality of life among patients with uterine fibroids, was designed in 2002s by James B et.al.
  Consisting of eight symptom items and twenty-nine health-related quality of life (HRQL) items of six subscales (concern, activities, energy/mood, control, self-consciousness, and sexual functioning), UFS-QOL is scored with a 5-point scale which demonstrates the patient' state of past 3 months. The final score (range, 0-100) is transformed based on a specific formula. Usually, a higher symptom severity score means more severe symptoms while a higher HRQL score indicates more perfect health
The degree of abdominal pain after myomectomy will be assessed by VAS（visual analogue scale, VAS） | through study completion, about June.2025
  VAS is the most commonly used one-dimensional measure of pain intensity. The scale consists mainly of a 100 mm straight line with one end indicating "completely painless" and the other end indicating "the most severe pain imaginable" or "extremely painful", etc. Patients will be asked to mark the line at the appropriate location to represent the intensity of the pain they are experiencing at the time
The blood loss will be assessed by PBLAC (Pictorial Blood Loss Assessment Chart (PBLAC) | through study completion, about June.2025
  The Pictorial Blood Loss Assessment Chart (PBLAC) proposed by Higham JM in 1990 is widely used internationally to evaluate menstrual flow. 1 Menstrual blood loss chart The menstrual blood loss chart is given different scores according to the different degrees of blood staining of each sanitary napkin: mild (1 point), the blood stained area < 1/3 of the whole sanitary napkin; Moderate (5 points): The blood stained area accounts for 1/3~3/5 of the whole sanitary napkin; Severe (20 points): The blood-stained area is basically the entire sanitary napkin.

CONTACTS AND LOCATIONS:
Overall Officials: Shixuan Wang, Phd, Study Chair — Huazhong University of Science and Technology
Locations (1):
- Shixuan Wang, Wuhan, None Selected, China

IPD SHARING:
Plan to Share IPD: No